CLINICAL TRIAL: NCT01266772
Title: The Effect of Montelukast on Anti-inflammatory Treatment and Asthma Exacerbation Prevention in Children Sensitive to Dust Mites.
Brief Title: Effect of Montelukast in Asthma in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Prof, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNN/213/10/KE; RNN/213/10/KE (Other: Medical University of Lodz)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Bronchial Asthma
Keywords: asthma; children; montelukast; treatment; exacerbation
MeSH Terms: conditions — Asthma | interventions — montelukast; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- montelukast group (Active Comparator): Children with asthma treated with montelukast and budesonide.
  Interventions: Drug: Montelukast sodium.
- Placebo group (Placebo Comparator): Children with asthma treated with placebo tablet and budesonide.
  Interventions: Drug: Placebo tablet and budesonide

INTERVENTIONS:
Drug: Montelukast sodium. — Children with asthma treated with montelukast and budesonide.
  Other Names: Montelukast and Budesonide
  Arms: montelukast group
Drug: Placebo tablet and budesonide — Children with asthma treated with placebo tablet and budesonide.
  Other Names: Placebo tablet and Budesonide.
  Arms: Placebo group

SUMMARY:
This is 9 month, placebo-controlled, double blind, randomised trial using the oral leucotrienes receptor antagonist montelukast (5 mg) in 160 children with mild and moderate asthma age 6-14 year old, sensitive to house dust mite. There are two study groups: montelukast group 80 patients and placebo group 80 patients. All patients will receive budesonide in dose sufficient to control asthma symptoms and short-acting beta agonist as needed. Medication used in the study: montelukast 5mg, budesonide. There are 7 doctor's visits - one initial visit (June) and 6 follow-up visits. First visit is on the first day of asthma symptom and each follow-up visit is every 6 weeks. Children with full asthma control (as measured by exhaled NO) had administered 100 mcg lower dose of budesonide and children with not fully control asthma had administered 100 mcg higher dose of budesonide.

DETAILED DESCRIPTION:
The most potent anti-inflammatory drugs in asthma are glucocorticosteroids. Corticosteroids, however have side effects and do not fully suppress the production or release of all inflammatory mediators. Amongst those less affected are cysteinyl leucotrienes, which are known to play a key role in asthma. Antileucotrienes have a bronchodilator and bronchoprotective potential and have thus became part of current treatment recommendations in asthma.

Owing to the beneficial effects of antileucotrienes and the efforts to keep steroid doses low, our study address the extent to which inhaled corticosteroids might be substituted or supplemented by these drugs. We used symptoms, frequency of exacerbation, exercise induced bronchoconstriction test, and exhaled NO during a stepwise reduction of steroid doses to assess the association between these variables and their relation to the patients' clinical benefit; we used airway hyperresponsiveness to assess inflammatory process in airways.

This is 9 month, placebo-controlled, double blind, randomised trial using the oral leucotrienes receptor antagonist montelukast (5 mg) in 160 children with mild and moderate asthma age 6-14 year old, sensitive to house dust mite. There are two study groups: montelukast group 80 patients and placebo group 80 patients. All patients will receive budesonide in dose sufficient to control asthma symptoms and short-acting beta agonist as needed. Medication used in the study: montelukast 5mg, budesonide. There are 7 doctor's visits - one initial visit (June) and 6 follow-up visits. First visit is on the first day of asthma symptom and each follow-up visit is every 6 weeks. Children with full asthma control (as measured by exhaled NO) had administered 100 mcg lower dose of budesonide and children with not fully control asthma had administered 100 mcg higher dose of budesonide.

Methods used in the study:

* doctor's exam
* asthma symptoms questionaire
* exhaled NO
* spirometry
* exercise induced bronchoconstriction test
* airway hyperresponsiveness test

End points:

* steroid doses sufficient to control asthma symptoms
* medium steroid dose/day times 6 month
* number of asthma exacerbations in 9 month period
* maximum fall of FEV1 in exercise induced bronchoconstriction test
* asthma symptoms scale and lung function
* number of patients with positive airway hyperresponsiveness test

ELIGIBILITY:
Inclusion Criteria:

* Children with bronchial asthma

Exclusion Criteria:

* All other serious diseases

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Steroid dose,medium steroid dose/day,number of asthma exacerbations,maximum fall of FEV1 in exercise, asthma symptoms, lung function, number of patients with positive airway hyperresponsiveness | 9 months
  * steroid doses sufficient to control asthma symptoms
  * medium steroid dose/day times 6 month
  * number of asthma exacerbations in 9 month period
  * maximum fall of FEV1 in exercise induced bronchoconstriction test
  * asthma symptoms scale and lung function
  * number of patients with positive airway hyperresponsiveness test

CONTACTS AND LOCATIONS:
Overall Officials: Agata Ożarek-Hanc, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland.; Iwona Stelmach, Prof., Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland

REFERENCES:
- [Derived] Stelmach I, Ozarek-Hanc A, Zaczeniuk M, Stelmach W, Smejda K, Majak P, Jerzynska J, Anna J. Do children with stable asthma benefit from addition of montelukast to inhaled corticosteroids: randomized, placebo controlled trial. Pulm Pharmacol Ther. 2015 Apr;31:42-8. doi: 10.1016/j.pupt.2015.01.004. Epub 2015 Jan 30. PMID 25640020